CLINICAL TRIAL: NCT03487302
Title: Assessment of White Matter Hyperintensities Burden in Adult Patients With Cyanotic Congenital Heart Disease: a Pilot Study
Brief Title: White Matter Hyperintensities Burden in Adult Patients With Cyanotic Congenital Heart Disease: a Pilot Study
Status: Completed | Type: Observational
Sponsor: IRCCS Policlinico S. Donato (Other)
Responsible Party: Principal Investigator, Francesco Sardanelli, Principal Investigator, IRCCS Policlinico S. Donato
Other Study IDs: LEUCO
Record Dates: First submitted 2018-03-20; First posted 2018-04-04 (Actual); Last update posted 2022-09-13 (Actual); Status verified 2022-09

CONDITIONS: Aging, Premature; Congenital Heart Disease; White Matter Hyperintensities
MeSH Terms: conditions — Aging, Premature; Heart Defects, Congenital

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- cCHD
  Interventions: Other: Brain MRI; Other: Neuropsychological test battery
- CONTROLS
  Interventions: Other: Brain MRI

INTERVENTIONS:
Other: Brain MRI — Acquisition of 3D T1-weighted, 3D FLAIR and GRE brain MRI scans
Other: Neuropsychological test battery — 1. Mini Mental State Examination (MMSE), Measso et al. (1993);
  2. Frontal Assessment Battery (FAB), Appollonio et al. (2005);
  3. Symbol Digit Test, Amodio et al. (2002);
  4. Digit Cancellation Test, Della Sala et al. (1992);
  5. Trial Making Test (TMT A-B), Giovagnoli et al. (1996);
  6. Weigl's Sorting Test, Laicona et al. (2000) and Inzaghi (2010);
  7. Digit Span, Orsini et al (1987);
  8. Corsi block-tapping test, Orsini et al. (1987);
  9. Babcock story recall test, Carlesimo et al. (2002);
  10. Phonemic verbal fluency in MDB, Caltagirone and Carlesimo (2010);
  11. Semantic verbal fluency, Novelli (1986);
  12. Imitating gestures, De Renzi et al. (1980);
  13. Coloured Progressive Matrices (CPM47), Measso et al. (1993).
  Groups: cCHD

SUMMARY:
The study aims at investigating the role of cyanotic congenital heart disease (cCHD) on brain aging. The investigators assume that due to congenital and acquired cardiovascular abnormalities, cCHD patients could show radiologic (and clinical) signs of precocious brain aging and eventual cognitive decline.

DETAILED DESCRIPTION:
White matter hyperintensities burden will be quantified through a semi-autamated software (ITK-SNAP)

ELIGIBILITY:
Inclusion Criteria:

* for the patient group, being an adult subject affected with cyanotic congenital heart disease, whether surgically corrected or not.
* for the control group, being an healthy subject.

Exclusion Criteria:

* any contraindication to magnetic resonance imaging;
* any pathological condition and/or symptomp that could alter the white matter hyperintensities burden, among which:

  * inflammatory, infectious, demyelinating or dysmyelinating diseases of the CNS;
  * ischemic, haemorrhagic or traumatic brain events and eventual gliotic and malacic or lacunar sequelae;
  * genetic diseases (whether mendelian or mitochondrial) of the CNS;
  * cerebral amyloid angiopathy;
  * CADASIL;
  * cerebral arteriovenous malformations;
  * primary or metastatic brain neoplasms which cause neurological symptoms and/or brain parenchymal sequelae from surgical excision;
  * patent oval foramen;
  * being pregnant;
  * migraine with aura (Bashir, Lipton, Ashina, & Ashina, 2013).

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: * for the patient group, being an adult subject affected with cyanotic congenital heart disease, whether surgically corrected or not;
  * for the control group, being an healthy subject.
Sampling Method: Probability Sample
Enrollment: 146 (Actual)
Dates: Start 2017-10-17 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
White matter hyperintensities volume expressed in mm^3 | 3 years
  Semi-automated quantification performed through ITK-SNAP

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Sardanelli, MD, Principal Investigator — IRCCS Policlinico S. Donato
Locations (1):
- IRCCS Policlinico San Donato, San Donato Milanese, Milano, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yushkevich PA, Piven J, Hazlett HC, Smith RG, Ho S, Gee JC, Gerig G. User-guided 3D active contour segmentation of anatomical structures: significantly improved efficiency and reliability. Neuroimage. 2006 Jul 1;31(3):1116-28. doi: 10.1016/j.neuroimage.2006.01.015. Epub 2006 Mar 20. PMID 16545965